CLINICAL TRIAL: NCT05992909
Title: Prophylactic Lymphovenous Bypass Procedure Following Inguinal Lymphadenectomy: A Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0203; NCI-2023-06282 (Other: NCI-Clinical Trials Registry)
Record Dates: First submitted 2023-08-04; First posted 2023-08-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Lymphadenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lymphovenous bypass procedure (LBP): A surgical procedure for treating lymphedema called lymphovenous bypass procedure (LBP), but it is usually only done after a patient develops lymphedema
  Interventions: Procedure: Lymphovenous bypass procedure

INTERVENTIONS:
Procedure: Lymphovenous bypass procedure — Participants will return to the clinic 14 days, 6 months, 12 months, 18 months, and 24 months after your surgery for measurements of your legs to see if there are changes over time

SUMMARY:
To learn if LBP can help to prevent lymphedema when it is performed at the time of surgery rather than after a patient has already developed the disease.

DETAILED DESCRIPTION:
Primary Objectives:

The objective of this study is to evaluate the protective benefit to performing LVB surgery at the time of ILND. In the secondary objective, we will compare the medical outcomes for patients that received the LVB surgery with those receiving standard surgery in whom the intervention could not be performed.

ELIGIBILITY:
Eligibility Criteria:

1. Patients greater than or equal to 18 years of age.
2. Patients willing to participate.
3. Patients able to complete informed consent.
4. Patients undergoing ILND.

Exclusion Criteria:

1. Patients taking anticoagulants within 7 days prior to surgery.
2. Patients that are known to be pregnant at the time of surgery.
3. Patients are available for follow-up less than 18 months or do not undergo measurements within the scheduled period.
4. Patients with BMI greater than 50.0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.03 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ashleigh Francis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org